CLINICAL TRIAL: NCT04478422
Title: Effects of a Muscle Training Program With and Without Vascular Occlusion in Pain, Functionality, Postural Control and Muscular Recruitment of Women With Patellophemoral Pain Syndrome: A Random Clinical Trial
Brief Title: Muscle Training With and Without Vascular Occlusion of Women With Patellofemoral Pain Syndrome: A Random Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiane Macedo (Other)
Responsible Party: Sponsor-Investigator, Christiane Macedo, Principal Investigator, Universidade Estadual de Londrina
Organization: Universidade Estadual de Londrina (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Vascular Occlusion in PFPS
Record Dates: First submitted 2020-07-10; First posted 2020-07-20 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Patellofemoral Pain Syndrome; Vascular Occlusion
Keywords: Patellofemoral Pain Syndrome; Partial Vascular Occlusion; Postural Balance; Electromyography; Physical Therapy.
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle strengthening with vascular occlusion (Experimental): Quadriceps strengthening exercises will be performed in isometric, concentric and eccentric phases, with partial occlusion to blood flow. The occlusion equipment will be positioned over the proximal portion of the lower limb to be treated, just below the gluteal fold and inguinal ligament (Tennent et al. 2017). The pressure must be maintained during all series of exercises (approximately 5 minutes) (Bryk et al. 2016; Ferraz et al. 2018; Giles et al. 2017).
  Interventions: Other: Muscle strengthening with vascular occlusion
- Conventional muscle strengthening (Active Comparator): Conventional quadriceps strengthening exercises will be performed in isometric, concentric and eccentric phases, without occlusion to blood flow.
  Interventions: Other: Conventional muscle strengthening

INTERVENTIONS:
Other: Muscle strengthening with vascular occlusion — The muscle strengthening group with partial vascular occlusion will perform the strengthening exercises: single leg squat on 25 ° inclined plane, eccentric + isometric + concentric quadriceps exercise and deep squat. The equipment for vascular occlusion will be positioned over the proximal portion of the lower limb to be treated, just below the gluteal fold and inguinal ligament (Tennent et al. 2017). The pressure must be maintained during all series of exercises (approximately 5 minutes) (Bryk et al. 2016; Ferraz et al. 2018; Giles et al. 2017). If necessary, the pressure can be adjusted at intervals and after the end of the exercise, an interval of 5 minutes is suggested for blood reperfusion.
  Arms: Muscle strengthening with vascular occlusion
Other: Conventional muscle strengthening — The conventional muscle strengthening group perform the same exercises as the intervention group: One-legged squat on a 25 ° inclined plane, eccentric + isometric + concentric quadriceps exercise and deep squat, however, without restriction on blood flow.
  Arms: Conventional muscle strengthening

SUMMARY:
Introduction: The treatment of Patellofemoral Pain Syndrome (PFPS) uses the strengthening of the knee and hip muscles. Studies propose the use of partial vascular occlusion (OVP) of the quadriceps muscle to increase muscle strength and endurance, without joint overload or discomfort to the patient. However, there is no consensus on the use in individuals with PFPS. Objective: To establish the effect of quadriceps muscle strengthening with OVP and low resistance to exercise on pain, functionality, postural control and muscle recruitment in women with patellofemoral dysfunction. Methods: Women with PFPS (n = 20) will respond to pain and functionality scales. The postural control and muscle recruitment of the quadriceps will also be evaluated in dynamic activities of single-legged squat and up / down stairs using a force platform and surface electromyography. After the initial assessment, the participants will be randomized into two groups: conventional quadriceps strengthening with greater resistance loads to exercise and quadriceps strengthening with OVP and low loads. And they will perform a six-week treatment protocol with exercises to strengthen the quadriceps. At the end of the intervention protocols, all of them will be reassessed immediately, after four and eight weeks. Expected Results: It is expected that the group submitted to exercises with OVP and lower load will present the same results of postural control and muscle recruitment compared to the conventional strengthening group. These results will indicate the possibility of using exercises and loads with less joint impairment.

ELIGIBILITY:
Inclusion Criteria:

Insidious onset of symptoms unrelated to trauma, pain for at least three months; pain greater than three (3/10) in at least three of the functional activities (squatting for a long time, going up or down stairs, kneeling, running, remaining in a sitting position for a long time), maximum 86 points on the Anterior Knee Pain Scale (AKPS).

Exclusion Criteria:

Signs and symptoms of other coexisting knee pathologies (arthrosis, prostheses, meniscal and ligament injuries), pain in other joints of the lower limb; lumbar spine pain, neurological, rheumatological, vascular and metabolic diseases; pregnancy; history of lower limb surgery; corticosteroid injection in the knee applied in the last three months, physiotherapy for knee rehabilitation in the last six months.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Pain in the knee by scale score | pre-intervention, immediately after, after four weeks
  Through Visual Analog Scale (VAS). The score ranges from 0 to 10, the higher the score, the greater the pain.
Change in functional capacity by scale score | pre-intervention, immediately after, after four weeks
  Using the Anterior Knee Pain Scale. The score ranges from 0 to 100, the higher the score, the better the functional capacity.
Change in functional capacity by scale score | pre-intervention, immediately after, after four weeks
  Using the Lysholm questionnaires. The score ranges from 0 to 100, the higher the score, the better the functional capacity.

SECONDARY OUTCOMES:
Change in Muscle activition by electromyography variables | pre-intervention, immediately after, after four weeks
  Muscle activition by surface electromyography of the quadriceps will be evaluated during one-legged squat activity and up and down stairs.
Change in quadriceps muscle strength | pre-intervention, immediately after, after four weeks
  Change in quadriceps muscle strength by portable dynamometry
Change in Postural control by pressure center variables | pre-intervention, immediately after, after four weeks
  Evaluation of postural control using a force platform will be evaluated during one-legged squat activity and up and down stairs.

CONTACTS AND LOCATIONS:
Locations (1):
- State University of Londrina, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tennent DJ, Hylden CM, Johnson AE, Burns TC, Wilken JM, Owens JG. Blood Flow Restriction Training After Knee Arthroscopy: A Randomized Controlled Pilot Study. Clin J Sport Med. 2017 May;27(3):245-252. doi: 10.1097/JSM.0000000000000377. PMID 27749358
- [Background] Bryk FF, Dos Reis AC, Fingerhut D, Araujo T, Schutzer M, Cury Rde P, Duarte A Jr, Fukuda TY. Exercises with partial vascular occlusion in patients with knee osteoarthritis: a randomized clinical trial. Knee Surg Sports Traumatol Arthrosc. 2016 May;24(5):1580-6. doi: 10.1007/s00167-016-4064-7. Epub 2016 Mar 12. PMID 26971109
- [Background] Ferraz RB, Gualano B, Rodrigues R, Kurimori CO, Fuller R, Lima FR, DE Sa-Pinto AL, Roschel H. Benefits of Resistance Training with Blood Flow Restriction in Knee Osteoarthritis. Med Sci Sports Exerc. 2018 May;50(5):897-905. doi: 10.1249/MSS.0000000000001530. PMID 29266093
- [Background] Giles LS, Webster KE, McClelland JA, Cook J. Does quadriceps atrophy exist in individuals with patellofemoral pain? A systematic literature review with meta-analysis. J Orthop Sports Phys Ther. 2013 Nov;43(11):766-76. doi: 10.2519/jospt.2013.4833. Epub 2013 Sep 9. PMID 24175596
- [Background] Thijs KM, Zwerver J, Backx FJ, Steeneken V, Rayer S, Groenenboom P, Moen MH. Effectiveness of Shockwave Treatment Combined With Eccentric Training for Patellar Tendinopathy: A Double-Blinded Randomized Study. Clin J Sport Med. 2017 Mar;27(2):89-96. doi: 10.1097/JSM.0000000000000332. PMID 27347857